CLINICAL TRIAL: NCT03555877
Title: Anti-hormonal Maintenance Treatment With the CDK4/6 Inhibitor Ribociclib After 1st Line Chemotherapy in Hormone Receptor Positive / HER2 Negative Metastatic Breast Cancer: A Phase II Trial
Brief Title: Anti-hormonal Therapie With Ribociclib in HR-positive / HER2- Negative Metastatic Breast Cancer
Acronym: AMICA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 97
Record Dates: First submitted 2018-02-16; First posted 2018-06-14 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer Metastatic
Keywords: Ribociclib; Anti-hormonal maintainance treatment; HR-positive; HER2-negative
MeSH Terms: interventions — ribociclib; Anastrozole; Letrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-hormonal treatment + ribociclib (Experimental): In the experimental arm ribociclib will be dosed on a flat scale of 600mg/day (corresponding to three 200mg tablets once daily, 3 week on, one week off). Anti-hormonal/endocrine treatment of choice of investigator: anastrozole, exemestane, letrozole, fulvestrant.
  Interventions: Drug: Ribociclib; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant
- Anti-hormonal treatment (Active Comparator): In the control arm patients will receive endocrine treatment only (of choise of investigator). Anti-hormonal/endocrine treatment of choice of investigator: anastrozole, exemestane, letrozole, fulvestrant.
  Interventions: Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: Ribociclib — Ribociclib in addition to endocrine maintenance therapy. Endocrine therapy, at the discretion of the investigator, could have already been started up to 4 weeks before randomization but not later than with first dose of ribociclib.
  Other Names: Kisqali
  Arms: Anti-hormonal treatment + ribociclib
Drug: Anastrozole — 1mg once daily as indicated in the SmPC
  Other Names: All marketed medicinal products with this active ingredient.
Drug: Letrozole — 2,5mg once daily as indicated in the SmPC
  Other Names: All marketed medicinal products with this active ingredient.
Drug: Exemestane — 25mg once daily as indicated in the SmPC
  Other Names: All marketed medicinal products with this active ingredient.
Drug: Fulvestrant — (prefilled syringes with fulvestrant 250mg each), 500mg given once a month, with an additional 500mg dose given two weeks after the first dose as indicated in the SmPC
  Other Names: All marketed medicinal products with this active ingredient.

SUMMARY:
This is a multicenter, prospective, randomized, open-label, controlled phase II study to test the addition of the CDK4/6 inhibitor ribociclib to anti-hormonal treatment as maintenance therapy in patients with disease control (at least stable disease) after 1st line chemotherapy.

DETAILED DESCRIPTION:
Although 1st line chemotherapy is effective in women with HR-positive HER2-negative breast cancer, PFS is usually around 6-8 months and 2nd or 3rd line treatments are by far less effective. Well tolerated maintenance treatments with the potential to prolong PFS and even OS are urgently needed. This study evaluates the impact of the addition of a CDK4/6 inhibitor to an anti-hormonal maintenance treatment of physicians´ choice.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Female patients.
3. Age ≥ 18 years old.
4. Histologically confirmed HER2-/HR+ locally advanced or metastatic invasive breast carcinoma assessed on the primary tumor and/or on the metastatic lesions (preferred).
5. Willingness and ability to provide archived formalin fixed paraffin embedded tissue block or a partial block from primary surgery and/or tumor or metastasis biopsy, which will be used for further breast cancer research.
6. Maintenance endocrine therapy could have already been started up to 6 weeks before randomization, but after achievement of tumor response or stable disease.
7. Maintenance therapy must be preceded prior to randomization by at least 4 cycles of a mono- or polychemotherapy. Tumor response or stable disease needs to be maintained to allow entry into the trial. Study treatment must start within 8 weeks of the last dose of chemotherapy.
8. Previous therapy with maximum one line of anti-hormonal treatment is allowed.
9. Previous neoadjuvant/adjuvant therapy is allowed. In case of cancer other than breast cancer, treatment should be completed more than 5 years before study entry.
10. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
11. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 4.03 Grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion).
12. The patient must be accessible for scheduled visits, treatment and follow-up. Patients registered on this trial must be treated at the participating center which could be the Principal or a Co- investigator's site.
13. Life-expectancy > 6 months.
14. The subjects need to be either A) of non-childbearing potential (documented postmenopausal or post hysterectomy) or B) childbearing potential with negative urinary pregnancy test (in this case patients need to use highly effective non-hormonal contraceptive).

Exclusion Criteria:

1. Uncontrolled/untreated central nervous system lesions.
2. Known severe hypersensitivity reactions to compounds similar to one of the investigational (active substance or peanut, soya or other excipients) and supportive treatment.
3. Inadequate organ function immediate prior to randomization including:

   * Hemoglobin < 10 g/dL
   * Absolute neutrophil count (ANC) < 2000/mm³ (< 2.0 x 109/L)
   * Platelets < 100,000/mm³ (< 100 x 109/L)
   * Alanine aminotransferase (ALAT/SGPT) and/or aspartate aminotransferase (ASAT/SGOT) > 2.0 x upper normal limits (ULN). If the patient has liver metastases, ALT and AST should not be ≥5 ULN.
   * Alkaline phosphatase (ALP) > 2.5 x ULN
   * Total serum bilirubin > 1.5 x ULN
   * Serum creatinine >1.5 x ULN or estimated creatinine clearance < 60 mL/min as calculated using the method standard for the Institution
4. Severe and relevant comorbidity that would interact with the participation in the study.
5. Previous malignant disease being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
6. Evidence for active infection including wound infections and anamnestic HIV or hepatitis.
7. QTc >450 msec or a family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes.
8. Uncontrolled electrolyte disorders that can compound the effects of a QTc prolonging drug (i.e. hypocalcemia, hypokalemia, hypomagnesemia).
9. Any of the following within 6 months prior to randomization: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE version 4.03 grade ≥ 2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
10. Other severe acute, uncontrolled or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
11. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
12. Patients treated within the last 7 days prior to randomization with drugs known to be CYP3A4 inhibitors or inducers (see section 11.4) or drugs that are known to prolong the QT interval.
13. Pregnant and lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Locally-assessed progression-free survival (PFS) | Up to 39 months
  Primary efficacy endpoint is locally-assessed progression-free survival (PFS) defined as the time elapsed between randomization and tumor progression or death from any cause.

SECONDARY OUTCOMES:
The impact on overall survival | Up to 39 months
  Overall survival (OS) defined as the time elapsed between treatment randomization and death from any cause
The clinical benefit rate | Up to 39 months
  Clinical benefit rate (CBR) defined as the proportion of subjects with best response of complete response, partial response, or stable disease for at least 24 weeks
Patient reported outcomes | Up to 39 months
  will be assessed using the General Quality of Life questionnaire (FACT-B), which will be filled in at study entry and every three month thereafter.
Number of participants with adverse events, serious adverse events and adverse events of special interest as assessed by CTCAE v4.03. | Up to 33 months
  Number of participants with adverse events, serious adverse events and adverse events of special interest as assessed by CTCAE v4.03 compared between the two treatment-arms.
The number of patients who reduced, interrupted or permanently discontinued treatment and the reasons for that. | Up to 33 months
  The number of patients who reduced, interrupted or permanently discontinued treatment and the reasons for that compared between two treatment-arms.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Decker, Prof. Dr., Principal Investigator — Gemeinschaftspraxis Onkologie Ravensburg
Locations (1):
- Studienzentrum Onkologie Ravensburg, Ravensburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gligorov J, Doval D, Bines J, Alba E, Cortes P, Pierga JY, Gupta V, Costa R, Srock S, de Ducla S, Freudensprung U, Mustacchi G. Maintenance capecitabine and bevacizumab versus bevacizumab alone after initial first-line bevacizumab and docetaxel for patients with HER2-negative metastatic breast cancer (IMELDA): a randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1351-60. doi: 10.1016/S1470-2045(14)70444-9. Epub 2014 Sep 28. PMID 25273343
- [Derived] Decker T, Ludtke-Heckenkamp K, Melnichuk L, Hirmas N, Lubbe K, Zahn MO, Schmidt M, Denkert C, Lorenz R, Muller V, Zahm DM, Mundhenke C, Bauer S, Thill M, Seropian P, Filmann N, Loibl S. Anti-hormonal maintenance treatment with the CDK4/6 inhibitor ribociclib after 1st line chemotherapy in hormone receptor positive / HER2 negative metastatic breast cancer: A phase II trial (AMICA). Breast. 2023 Dec;72:103575. doi: 10.1016/j.breast.2023.08.007. Epub 2023 Sep 1. PMID 37690320
- See also: GBG website active studies — http://www.gbg.de/de/studien/aktive-studien.php